CLINICAL TRIAL: NCT06028711
Title: The Impact of Education on the Rehabilitation of Patients Hospitalized Due to Chronic Obstructive Pulmonary Disease.
Brief Title: Education Impact on Rehabilitation of Hospitalized Patients with Chronic Obstructive Pulmonary Disease.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Renata Borys, Principal Investigator, University of Rzeszow
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: URzeszow/2023/06/0034/W
Record Dates: First submitted 2023-08-25; First posted 2023-09-08 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: pulmonary rehabilitation; COPD patients' education
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: random selection to two groups (study group and control group)
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Education program and Pulmonary rehabilitation (Experimental): Conventional pulmonary rehabilitation coupled with original education program.
  Interventions: Other: Education program; Other: Pulmonary rehabilitation
- Pulmonary rehabilitation (Other): Conventional pulmonary rehabilitation
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Education program — Patients in a study group will participate in daily education program using an original brochure containing information on the benefits of appropriately adapted physical activity, practical tips on airway clearance techniques or physical exercise, and risk factors for exacerbation of COPD.
  Arms: Education program and Pulmonary rehabilitation
Other: Pulmonary rehabilitation — The patients will participate in a 14-day rehabilitation program (Monday to Saturday). Treatments and therapies will be continued for a maximum of two hours daily. The program will be applied individually to each patient and include active and assisted exercises, effective cough exercises, pursed-lips breathing, positive expiratory pressure exercises, exercises to strengthen the diaphragm and intercostal muscles and cardiopulmonary exercises.

SUMMARY:
The planned research will enable the assessment of rehabilitation's effects using two pulmonary rehabilitation models: conventional and supplemented with an education program for patients hospitalized due to chronic obstructive pulmonary disease.

DETAILED DESCRIPTION:
The planned group size is 100 patients diagnosed with chronic obstructive pulmonary disease (COPD) and hospitalized due to exacerbation. The given population was calculated based on the sampling calculator, considering the following parameters: fraction size, confidence level, and maximum error.

Eligible patients will be randomly divided into two groups: a study group (50 patients) undergoing pulmonary rehabilitation supplemented with an education program and a control group (50 patients) undergoing conventional pulmonary rehabilitation.

Patients of both groups will be included in a 14-day rehabilitation program (Monday to Saturday). Treatments and therapies will be continued for a maximum of two hours daily. The program will be applied individually to each patient, including active and assisted exercises, effective cough exercises, pursed-lips breathing, positive expiratory pressure exercises, exercises to strengthen the diaphragm and intercostal muscles, and cardiopulmonary exercises. Patients from the study group will additionally undergo daily education using an original brochure containing information on the benefits of appropriately adapted physical activity, practical tips on airway clearance techniques or physical exercise, and risk factors for exacerbation of COPD.

The test will be performed three times: before the start of rehabilitation, after completing the rehabilitation program, and the follow-up after two months from the end of hospitalization to assess long-term effects. After the end of the study, people from the control group will also undergo education.

The patients' condition and the rehabilitation effects will be assessed using the following measures:

* Dynamic lung capacities (spirometry)
* Oxygen saturation and pulse rate (pulse oximeter)
* Acid-base balance (gasometry)
* Exercise tolerance (6-minute walking test)
* Fatigue (modified Borg scale)
* Physical performance (Fullerton functional fitness test)
* Dyspnea assessment (MRC dyspnea scale)
* Quality of life (WHOQOL-BREF)
* Anxiety and depression (HADS scale)
* Activities of daily living (Lawton IADL scale)

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed chronic obstructive pulmonary disease in the exacerbation phase
* Moderate stage (II) of the disease
* Independence in basic activities of daily living (above 86 points on the Barthel scale)
* Age 55 y.o. to 70 y.o.
* No additional respiratory support (e.a. cardiopulmonary bypass machine, ventilator)
* Informed, voluntary consent to participate in research.

Exclusion Criteria:

* Diagnosed chronic obstructive pulmonary disease in remission
* Stages I, III and IV of the disease - a forms with mild, severe, and very severe obstruction
* Hospitalization in the intensive care unit, current health condition precluding participation in the study
* Age under 55 y.o. and over 70 y.o.
* Cognitive deficits impairing the ability to understand and execute commands
* Concomitant oncological, neurological, orthopedic, and psychiatric diseases may affect the examined persons' circulatory and respiratory functions, functional efficiency, quality of life, and emotional state.
* Failure to complete a 14-day rehabilitation program
* Lack of informed, voluntary consent to participate in research.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-07-28 (Actual); Primary Completion 2024-09-02 (Actual); Study Completion 2024-10-07 (Actual)

PRIMARY OUTCOMES:
Dynamic lung capacities (spirometry) | First examination- before the start of the interventions
  Measurements will be performed with certified spirometer and the parameters analyzed will be Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 Second (FEV1) measured in litres [L].
Dynamic lung capacities (spirometry) | Second examination- at the end of the 14-day rehabilitation program
  Measurements will be performed with certified spirometer and the parameters analyzed will be Forced Vital Capacity (FVC) and Forced Expiratory Volume in 1 Second (FEV1) measured in litres [L].
Modified Tiffeneau-Pinelli index (spirometry) | First examination- before the start of the interventions
  Measurement will be performed with certified spirometer and the parameter analyzed will be the ratio of Forced Expiratory Volume in 1 Second to Forced Vital Capacity (FEV1/FVC ratio) presented as a decimal fraction.
Modified Tiffeneau-Pinelli index (spirometry) | Second examination- at the end of the 14-day rehabilitation program
  Measurement will be performed with certified spirometer and the parameter analyzed will be the ratio of Forced Expiratory Volume in 1 Second to Forced Vital Capacity (FEV1/FVC ratio) presented as a decimal fraction.
Oxygen saturation | First examination- before the start of the interventions
  Measurements will be performed with pulse oximeter and the parameter analyzed will be oxygen saturation by pulse oximetry (SpO2, percentage of oxygen in patients' blood).
Oxygen saturation | Second examination- at the end of the 14-day rehabilitation program
  Measurements will be performed with pulse oximeter and the parameter analyzed will be oxygen saturation by pulse oximetry (SpO2, percentage of oxygen in patients' blood).
Pulse rate | First examination- before the start of the interventions
  Measurements will be performed with pulse oximeter and the parameter analyzed will be the number of patients' heart beats per minute.
Pulse rate | Second examination- at the end of the 14-day rehabilitation program
  Measurements will be performed with pulse oximeter and the parameter analyzed will be the number of patients' heart beats per minute.
Acid-base balance | First examination- before the start of the interventions
  The gasometry results will be taken from patients' medical documentation. The parameters analyzed will be oxygen pressure (pO2) and carbon dioxide pressure (pCO2).
Acid-base balance | Second examination- at the end of the 14-day rehabilitation program
  The gasometry results will be taken from patients' medical documentation. The parameters analyzed will be oxygen pressure (pO2) and carbon dioxide pressure (pCO2).
Exercise tolerance assessed by 6-minute walking test (6MWT) | First examination- before the start of the interventions
  The test will be performed in 20-meter long hospital corridor. The patient should walk the distance at his own rhythm and pace, using orthopedic aids (if necessary). The patient will be informed that they can stop the test at any time if they feel it is necessary. The distance traveled in meters in 6 minutes will be analyzed.
Exercise tolerance assessed by 6-minute walking test (6MWT) | Second examination- at the end of the 14-day rehabilitation program
  The test will be performed in 20-meter long hospital corridor. The patient should walk the distance at his own rhythm and pace, using orthopedic aids (if necessary). The patient will be informed that they can stop the test at any time if they feel it is necessary. The distance traveled in meters in 6 minutes will be analyzed.
Physical performance assessment by Fullerton functional fitness test | First examination- before the start of the interventions
  The test comprising muscle endurance, aerobic capacity, flexibility, agility, and balance assessment. The test consist of 6 activities: 1. Arm Curl Test (number of forearm flexions in 30 seconds); 2. Back Scratch (the distance between middle fingers); 3. 30 Second Chair Stand (number of standings in 30 seconds); 4. Chair Sit-and-Reach ( '+' if fingers can reach toes in sitting position, '-' if fingers cannot reach toes in sitting position); 5. 8 - Foot Up-and-Go (8-foot walking time); 6. 2-Minute Step-in-Place (the number of lifts of the right leg).
Physical performance assessment by Fullerton functional fitness test | Second examination- at the end of the 14-day rehabilitation program
  The test comprising muscle endurance, aerobic capacity, flexibility, agility, and balance assessment. The test consist of 6 activities: 1. Arm Curl Test (number of forearm flexions in 30 seconds); 2. Back Scratch (the distance between middle fingers); 3. 30 Second Chair Stand (number of standings in 30 seconds); 4. Chair Sit-and-Reach ( '+' if fingers can reach toes in sitting position, '-' if fingers cannot reach toes in sitting position); 5. 8 - Foot Up-and-Go (8-foot walking time); 6. 2-Minute Step-in-Place (the number of lifts of the right leg).
Fatigue assessment using modified Borg scale | First examination- before the start of the interventions
  Fatigue will be examined during physical activity and the level of fatigue will be marked on a scale from 1 (no fatigue) to 10 (very very hard fatigue).
Fatigue assessment using modified Borg scale | Second examination- at the end of the 14-day rehabilitation program
  Fatigue will be examined during physical activity and the level of fatigue will be marked on a scale from 1 (no fatigue) to 10 (very very hard fatigue).
Fatigue assessment using modified Borg scale | Third examination - two months after discharge from the hospital (follow- up)
  Fatigue will be examined during physical activity and the level of fatigue will be marked on a scale from 1 (no fatigue) to 10 (very very hard fatigue).
Dyspnea assessment with Medical Research Council dyspnea scale | First examination- before the start of the interventions
  Perceived breathlessness degree will be marked on a scale 0 (no breathlessness) to 4 (breathlessness at rest).
Dyspnea assessment with Medical Research Council dyspnea scale | Second examination- at the end of the 14-day rehabilitation program
  Perceived breathlessness degree will be marked on a scale 0 (no breathlessness) to 4 (breathlessness at rest).
Dyspnea assessment with Medical Research Council dyspnea scale | Third examination - two months after discharge from the hospital (follow- up)
  Perceived breathlessness degree will be marked on a scale 0 (no breathlessness) to 4 (breathlessness at rest).
Quality of life assessment using World Health Organization Quality-of-Life Scale (WHOQOL-BREF) | First examination- before the start of the interventions
  Assessment of quality of life, health and other areas. The scale contains 26 items, divided into four domains: physical health (7 items), psychological health (6 items), social relations (3 items), and environmental health (8 items), as well overall quality of life and general health (2 items). Patients express how much they have experienced the items in the preceding 2 weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely). The final score is transformed linearly to a 0-100-scale, where higher scores denote higher quality of life.
Quality of life assessment using World Health Organization Quality-of-Life Scale (WHOQOL-BREF) | Second examination- at the end of the 14-day rehabilitation program
  Assessment of quality of life, health and other areas. The scale contains 26 items, divided into four domains: physical health (7 items), psychological health (6 items), social relations (3 items), and environmental health (8 items), as well overall quality of life and general health (2 items). Patients express how much they have experienced the items in the preceding 2 weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely). The final score is transformed linearly to a 0-100-scale, where higher scores denote higher quality of life.
Quality of life assessment using World Health Organization Quality-of-Life Scale (WHOQOL-BREF) | Third examination - two months after discharge from the hospital (follow- up)
  Assessment of quality of life, health and other areas. The scale contains 26 items, divided into four domains: physical health (7 items), psychological health (6 items), social relations (3 items), and environmental health (8 items), as well overall quality of life and general health (2 items). Patients express how much they have experienced the items in the preceding 2 weeks on a 5-point Likert scale ranging from 1 (not at all) to 5 (completely). The final score is transformed linearly to a 0-100-scale, where higher scores denote higher quality of life.
Anxiety and depression assessment using HADS scale | First examination- before the start of the interventions
  The scale consists of 16 statements to which the respondent refers on a four-point scale. Eight statements are used to measure anxiety and depression, each of which is rated on a scale of 0 to 3 points. The cut-off threshold is 7 points for depression and 7 points for anxiety. The intensity of depressed mood and anxiety will be analyzed.
Anxiety and depression assessment using HADS scale | Second examination- at the end of the 14-day rehabilitation program
  The scale consists of 16 statements to which the respondent refers on a four-point scale. Eight statements are used to measure anxiety and depression, each of which is rated on a scale of 0 to 3 points. The cut-off threshold is 7 points for depression and 7 points for anxiety. The intensity of depressed mood and anxiety will be analyzed.
Anxiety and depression assessment using HADS scale | Third examination - two months after discharge from the hospital (follow- up)
  The scale consists of 16 statements to which the respondent refers on a four-point scale. Eight statements are used to measure anxiety and depression, each of which is rated on a scale of 0 to 3 points. The cut-off threshold is 7 points for depression and 7 points for anxiety. The intensity of depressed mood and anxiety will be analyzed.
Activities of daily living assesment using Lawton Instrumental Activities of Daily Living (IADL) Scale | First examination- before the start of the interventions
  Life independence test, i.e. ensuring the functioning of the household by a sick person based on his/her ability to cope in the external environment or with a complex activity such as using the telephone and ensuring the related opportunities. The ability of basic functioning in the environment will be analyzed and each of 8 items will be rate trichotomously (1 = unable, 2 = needs assistance, 3 = independent) and sum the eight responses. The final total score ranges from 8 (low functioning, dependent) to 24 (high function, independent).
Activities of daily living assesment using Lawton Instrumental Activities of Daily Living (IADL) Scale | Second examination- at the end of the 14-day rehabilitation program
  Life independence test, i.e. ensuring the functioning of the household by a sick person based on his/her ability to cope in the external environment or with a complex activity such as using the telephone and ensuring the related opportunities. The ability of basic functioning in the environment will be analyzed and each of 8 items will be rate trichotomously (1 = unable, 2 = needs assistance, 3 = independent) and sum the eight responses. The final total score ranges from 8 (low functioning, dependent) to 24 (high function, independent).
Activities of daily living assesment using Lawton Instrumental Activities of Daily Living (IADL) Scale | Third examination - two months after discharge from the hospital (follow- up)
  Life independence test, i.e. ensuring the functioning of the household by a sick person based on his/her ability to cope in the external environment or with a complex activity such as using the telephone and ensuring the related opportunities. The ability of basic functioning in the environment will be analyzed and each of 8 items will be rate trichotomously (1 = unable, 2 = needs assistance, 3 = independent) and sum the eight responses. The final total score ranges from 8 (low functioning, dependent) to 24 (high function, independent).

CONTACTS AND LOCATIONS:
Overall Officials: Renata Borys, MSc, Principal Investigator — University of Rzeszow; Agnieszka Guzik, A/Prof., Study Director — University of Rzeszow; Magdalena Kołodziej, PhD, Study Chair — University of Rzeszow
Locations (1):
- University of Rzeszów, Rzeszów, Poland